CLINICAL TRIAL: NCT05965102
Title: A Prospective, Single-arm, Single-center, Exploratory Clinical Study of Tirelizumab Combined With Chemotherapy in First-line Treatment of ECOG PS 2 Points in Relapsed/Metastatic Non-small Cell Lung Cancer
Brief Title: Tirellizumab Combined With Chemotherapy Monotherapy for Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-ZF-10
Record Dates: First submitted 2023-04-23; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tirelizumab in combination with chemotherapy monotherapy (Experimental): This study is a one-arm, exploratory study and does not involve randomization. There was only one trial group of tirellizumab plus chemotherapy monotherapy.
  Interventions: Drug: Tirelizumab；Chemotherapy monotherapy

INTERVENTIONS:
Drug: Tirelizumab；Chemotherapy monotherapy — Tirelizumab combined with chemotherapy in first-line treatment of relapsed/metastatic non-small cell lung cancer with ECOG PS score of 2

SUMMARY:
This is a prospective, single-arm, single-center, exploratory clinical trial to evaluate the efficacy and safety of the PD-1 antibody tirelizumab combined with chemotherapy monotherapy in patients with relapsed/metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center, exploratory clinical trial to evaluate the efficacy and safety of the PD-1 antibody tirellizumab combined with chemotherapy monotherapy in patients with relapsed/metastatic non-small cell lung cancer. This study prospectively collected disease history, treatment history, demographic data, baseline data during treatment, each treatment visit data, efficacy data, and safety data of NSCLC patients with EGFR and ALK driver negative ECOG PS 2 scores treated with tirellizumab combined with monotherapy. The subjects did not voluntarily withdraw from the test or the researchers believed that the subjects were not suitable for further test. Each subject will be treated until the disease progresses or the toxic and side effects caused by the drugs are intolerable, and the follow-up treatment plan, treatment status and survival data of the patients still need to be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed recurrent/metastatic non-small cell lung cancer with local recurrence or distant metastasis after prior radiotherapy and/or surgery, or with distant metastasis at the time of admission.
2. The age range is between 18 and 85.
3. Predicted survival ≥12 weeks.

Exclusion Criteria:

1. Patients with other malignant tumors.
2. Positive tests for EGFR mutation and ALK fusion gene have been confirmed.
3. Partial comorbidity.
4. other.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Baseline C1D21 and C1D21 were followed by radiographic evaluations every 6 weeks (±7 days) until radiographic PD was recorded.
  Proportion of subjects assessed with CR or PR based on RECIST v1.1 criteria as a percentage of all enrolled patients

SECONDARY OUTCOMES:
Disease control rate | Baseline C1D21 and C1D21 were followed by radiographic evaluations every 6 weeks (±7 days) until radiographic PD was recorded.
  Proportion of subjects assessed as CR, PR, or SD based on RECIST v1.1 criteria.
Progression-free survival time | Baseline C1D21 and C1D21 were followed by radiographic evaluations every 6 weeks (±7 days) until radiographic PD was recorded.
  The time between the patient's first treatment date and any recorded tumor progression or death from any cause.
Overall survival time | Baseline C1D21 and C1D21 were followed by radiographic evaluations every 6 weeks (±7 days) until radiographic PD was recorded.
  The time between the patient's date of first treatment and death from any cause.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novello S, Le Chevalier T. Chemotherapy for non-small-cell lung cancer. Part 1: Early-stage disease. Oncology (Williston Park). 2003 Mar;17(3):357-64. PMID 12661267
- [Background] Langer CJ, Besse B, Gualberto A, Brambilla E, Soria JC. The evolving role of histology in the management of advanced non-small-cell lung cancer. J Clin Oncol. 2010 Dec 20;28(36):5311-20. doi: 10.1200/JCO.2010.28.8126. Epub 2010 Nov 15. PMID 21079145
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leal TA, Riess JW, Jensen E, Zhao B, Pietanza MC, Brahmer JR. Five-Year Outcomes With Pembrolizumab Versus Chemotherapy for Metastatic Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score >/= 50. J Clin Oncol. 2021 Jul 20;39(21):2339-2349. doi: 10.1200/JCO.21.00174. Epub 2021 Apr 19. PMID 33872070
- [Background] Zhou C, Chen G, Huang Y, Zhou J, Lin L, Feng J, Wang Z, Shu Y, Shi J, Hu Y, Wang Q, Cheng Y, Wu F, Chen J, Lin X, Wang Y, Huang J, Cui J, Cao L, Liu Y, Zhang Y, Pan Y, Zhao J, Wang L, Chang J, Chen Q, Ren X, Zhang W, Fan Y, He Z, Fang J, Gu K, Dong X, Zhang T, Shi W, Zou J; CameL Study Group. Camrelizumab plus carboplatin and pemetrexed versus chemotherapy alone in chemotherapy-naive patients with advanced non-squamous non-small-cell lung cancer (CameL): a randomised, open-label, multicentre, phase 3 trial. Lancet Respir Med. 2021 Mar;9(3):305-314. doi: 10.1016/S2213-2600(20)30365-9. Epub 2020 Dec 18. PMID 33347829
- [Background] Middleton G, Brock K, Savage J, Mant R, Summers Y, Connibear J, Shah R, Ottensmeier C, Shaw P, Lee SM, Popat S, Barrie C, Barone G, Billingham L. Pembrolizumab in patients with non-small-cell lung cancer of performance status 2 (PePS2): a single arm, phase 2 trial. Lancet Respir Med. 2020 Sep;8(9):895-904. doi: 10.1016/S2213-2600(20)30033-3. Epub 2020 Mar 19. PMID 32199466